CLINICAL TRIAL: NCT03022097
Title: A 24-week Treatment, Randomised, Parallel-group, Double Blinded, Double-Dummy, Multicenter Study to Assess the Efficacy and Safety of Aclidinium Bromide/Formoterol Fumarate Compared With Individual Components and Placebo and Aclidinium Bromide Compared With Placebo When Administered to Patients With Stable Chronic Obstructive Pulmonary Disease.
Brief Title: Study to Assess Efficacy and Safety of Aclidinium Bromide and Aclidinium Bromide/Formoterol Fumarate in Stabile COPD Patients
Acronym: AVANT
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: AstraZeneca (Industry)
Collaborators: Parexel (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: D6570C00002; M-AS464-30 (Other: Astrazenca)
Record Dates: First submitted 2017-01-13; First posted 2017-01-16 (Estimated); Results first posted 2025-03-26 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — aclidinium bromide; Formoterol Fumarate

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Experimental 1 (Experimental): Aclidinium bromide 400μg/Formoterol fumarate 12 μg
  Interventions: Drug: Aclidinium bromide/formoterol Fixed-Dose Combination
- Experimental 2 (Experimental): Aclidinium bromide 400 μg
  Interventions: Drug: Aclidinium bromide
- Comparator (Active Comparator): Formoterol fumarate 12 μg
  Interventions: Drug: Formoterol Fumarate
- Placebo (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aclidinium bromide/formoterol Fixed-Dose Combination — Inhaled Aclidinium bromide/formoterol Fixed-Dose Combination, twice per day via Genuair
  Arms: Experimental 1
Drug: Aclidinium bromide — Inhaled Aclidinium bromide 400 μg, twice per day via Genuair
  Arms: Experimental 2
Drug: Formoterol Fumarate — Inhaled Formoterol Fumarate 12 μg, twice per day via Turbuhaler
  Arms: Comparator
Drug: Placebo — Inhaled dose-matched placebo, twice per day via Genuair or via Turbuhaler
  Arms: Placebo

SUMMARY:
This is a multiple dose, randomised, parallel, double blind, double dummy, multicentre and multinational Phase III study to determine the efficacy and safety of Aclidinium bromide/Formoterol fumarate compared with individual components and placebo and Aclidinium bromide compared with Placebo when administered to patients with stable Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

* 1. Adult male or non-pregnant, non-lactating female patients aged ≥40
* 2. Patients with a diagnosis of COPD prior to Visit 1 (screening)
* 3. Patients with moderate to severe stable COPD (Stage II or Stage III) at Visit 1: post-bronchodilator FEV1 ≥30% and < 80% and post-bronchodilator FEV1/Forced vital capacity (FVC) < 70%
* 4. Current or former smokers with a smoking history of ≥ 10 pack-years
* 5. Patients able to perform repeatable pulmonary function testing for FEV1 according to the American Thoracic Society (ATS)/European Respiratory Society (ERS) 2005 criteria at Visit 1(screening)
* 6. Patients who understand the study procedures and are willing to participate in the study as indicated by signing the informed consent

Exclusion Criteria:

* 1. Involvement in the planning and/or conduct of the study (applies to AstraZeneca staff and/or site staff) or patients employed by or relatives of the employees of the site or sponsor.
* 2. Previous enrolment or randomisation in the present study
* 3. History or current diagnosis of asthma
* 4. Any respiratory tract infection (including the upper respiratory tract) or COPD exacerbation (including the mild COPD exacerbation) within 6 weeks prior to screening or during the run-in period
* 5. Patients hospitalized for COPD exacerbation (an emergency room visit for longer than 24 hours will be considered a hospitalization) within 3 months prior to screening and during the run-in period
* 6. Clinically significant respiratory conditions other than COPD
* 7. Patients who in the Investigator's opinion may need to start a pulmonary rehabilitation program during the study and/or patients who started/finished it within 3 months prior to screening
* 8. Use of long-term oxygen therapy (≥15 hours/day)
* 9. Patient who does not maintain regular day/night, waking/sleeping cycles including night shift workers
* 10. Clinically significant cardiovascular conditions
* 11. Patients with Type I or uncontrolled Type II diabetes, uncontrolled hypo-or hyperthyroidism, hypokalaemia, or hyperadrenergic state, uncontrolled or untreated hypertension
* 12. Patients with QT corrected interval (QTc) using Fridericia formula (QTcF) (QTc=QT/ Duration in milliseconds between two R peaks of two consecutive QRS complexes (RR1/3) >470 msec as indicated in the centralised reading report assessed at Screening (Visit 1)
* 13. Patients with clinically significant abnormalities in the clinical laboratory tests, ECG parameters (other than QTcF) or in the physical examination at Visit 1 (screening)
* 14. Patients with abnormal liver function tests defined as Aspartate aminotransferase (AST), Alanine aminotransferase (ALT), or total bilirubin ≥ 2.5 times upper limit of normal ranges at screening
* 15. Patient with known non-controlled history of infection with human immunodeficiency virus and/or active hepatitis
* 16. Patient with a history of hypersensitivity reaction to inhaled anticholinergic drugs, sympathomimetic amines, inhaled medication or any component thereof
* 17. Patient with known narrow-angle glaucoma, symptomatic bladder neck obstruction, acute urinary retention, or patients with symptomatic non-stable prostatic hypertrophy
* 18. History of malignancy of any organ system (including lung cancer), treated or untreated, within the past 5 years other than basal or squamous cell skin cancer
* 19. Any other serious or uncontrolled physical or mental dysfunction
* 20. Patients with a history (within 2 years prior to Visit 1 (screening) of drug and/or alcohol abuse that may prevent study compliance based on the Investigator judgment
* 21. Patients unlikely to be cooperative or cannot comply with the study procedures
* 22. Patients treated with any investigational drug within 30 days (or 6 half-lives, whichever is longer) prior to screening
* 23. Patients who intended to use any concomitant medication not permitted by this protocol or who had not undergone the required washout period for a particular prohibited medication
* 24. Patients unable to give consent, or patients of consenting age but under guardianship, or vulnerable patients
* 25. Any other conditions that, in the Investigator's opinion, might have indicated the patient to be unsuitable for the study

Ages: 40 Years to 130 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1625 (Actual)
Dates: Start 2017-02-02 (Actual); Primary Completion 2022-04-14 (Actual); Study Completion 2022-04-14 (Actual)

CONTACTS AND LOCATIONS:
Locations (52):
- China (33):
  - Research Site, Baotou
  - Research Site, Beijing
  - Research Site, Cangzhou
  - Research Site, Changchun
  - Research Site, Changsha
  - Research Site, Chengdu
  - Research Site, Guangzhou
  - Research Site, Haikou
  - Research Site, Hangzhou
  - Research Site, Hefei
  - Research Site, Hengyang
  - Research Site, Hohhot
  - Research Site, Liangyugang
  - Research Site, Linhai
  - Research Site, Nanchang
  - Research Site, Nanjing
  - Research Site, Qiqihar
  - Research Site, Shanghai
  - Research Site, Shanxi
  - Research Site, Shengyang
  - Research Site, Shenzhen
  - Research Site, Shijiazhuang
  - Research Site, Taiyuan
  - Research Site, Tianjin
  - Research Site, Wenzhou
  - Research Site, Wuxi
  - Research Site, Xi'an
  - Research Site, Xiamen
  - Research Site, Xining
  - Research Site, Yangzhou
  - Research Site, Yanji
  - Research Site, Yinchuan
  - Research Site, Zhanjiang
- India (10):
  - Research Site, Ahmedabad
  - Research Site, Alappuzha
  - Research Site, Ernākulam
  - Research Site, Guntur
  - Research Site, Jaipur
  - Research Site, Kozhikode
  - Research Site, Mysore
  - Research Site, Nagpur
  - Research Site, Pune
  - Research Site, Vijayawada
- Philippines (4):
  - Research Site, Caloocan
  - Research Site, Iloilo City
  - Research Site, Manila
  - Research Site, Quezon City
- Taiwan (3):
  - Research Site, Keelung
  - Research Site, Taichung
  - Research Site, Taipei
- Vietnam (2):
  - Research Site, Hanoi
  - Research Site, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers can request access to anonymized individual patient-level data from AstraZeneca group of companies sponsored clinical trials via the request portal. All request will be evaluated as per the AZ disclosure commitment: https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Supporting Information: Study Protocol, SAP
Time Frame: AstraZeneca will meet or exceed data availability as per the commitments made to the EFPIA Pharma Data Sharing Principles. For details of our timelines, please rerefer to our disclosure commitment at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
Access Criteria: When a request has been approved AstraZeneca will provide access to the de-identified individual patient-level data in an approved sponsored tool . Signed Data Sharing Agreement (non-negotiable contract for data accessors) must be in place before accessing requested information. Additionally, all users will need to accept the terms and conditions of the SAS MSE to gain access. For additional details, please review the Disclosure Statements at https://astrazenecagrouptrials.pharmacm.com/ST/Submission/Disclosure.
URL: https://astrazenecagroup-dt.pharmacm.com/DT/Home

REFERENCES:
- See also: CSR Synopsis — https://filehosting-v2.pharmacm.com/api/Attachment/Download?tenantId=80217111&parentIdentifier=D6570C00002&attachmentIdentifier=0136b8b2-5200-4274-bc73-a2b8e01690db&fileName=d6570c00002-CSR-synopsis.pdf&versionIdentifier=

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 81 study centers in 5 countries China(50), India (15), Philippines (8), Taiwan (3) and Vietnam (5) between 02 February 2017 and 14 April 2022
Pre-assignment Details: Subjects fulfilling inclusion/exclusion criteria at the time of the Screening entered into a run-in period of 14 ± 3 days to assess their disease stability before randomization. Participants who met the inclusion and none of the exclusion were considered for enrolment into the study. All study assessments were performed as per the schedule of assessments. A total of 1625 participants (consented) and undergone washout period and 1066 were randomised to treatment.
Groups:
- AB/FF 400/12 μg: Aclidinium bromide/formoterol fumarate fixed dose combination 400/12 μg
- AB 400 μg: Aclidinium bromide AB 400 μg
- FF 12 μg: Formoterol 12 μg
Period: Overall Study
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | Placebo
Started (Randomized Analysis Set) | 265 | 267 | 265 | 269
Received Treatment (Safety Analysis Set) | 263 | 266 | 264 | 269
Received Treatment With a Baseline FEV1 (Intention-to-Treat Analysis Set) | 262 | 265 | 259 | 267
Completed Treatment (Treatment completed if taken until Week 24.) | 243 | 247 | 230 | 230
Completed (Completed if treatment was taken until Week 24 or if treatment was discontinued early, but the subject was followed up in the study until Week 24.) | 244 | 248 | 233 | 235
Not Completed | 21 | 19 | 32 | 34
Not completed — Adverse Event | 3 | 4 | 1 | 3
Not completed — Progressive Disease | 2 | 0 | 5 | 2
Not completed — Lack of Efficacy | 0 | 0 | 3 | 3
Not completed — Protocol Violation | 1 | 0 | 1 | 0
Not completed — Withdrawal by Subject | 11 | 13 | 15 | 21
Not completed — Lost to Follow-up | 0 | 0 | 1 | 1
Not completed — Other | 4 | 1 | 6 | 4
Not completed — Due to COVID-19 pandemic | 0 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Safety population comprising all participants randomised to a treatment group who received at least one dose of double-blind investigational treatment (Safety Analysis Set).
Groups:
- Total: Total of all reporting groups
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | Placebo | Total
Number analyzed (Participants) | 263 | 266 | 264 | 269 | 1062
Age, Continuous [Mean (Standard Deviation); unit: Years] | 65.3 (7.1) | 65.4 (6.8) | 65.4 (7.6) | 64.9 (6.9) | 65.2 (7.1)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 256 | 254 | 251 | 256 | 1017
  Female | 7 | 12 | 13 | 13 | 45
Race (NIH/OMB) [Count of Participants; unit: Participants] — Race
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 263 | 266 | 264 | 269 | 1062
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 0 | 0 | 0 | 0 | 0
    White | 0 | 0 | 0 | 0 | 0
    More than one race | 0 | 0 | 0 | 0 | 0
    Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race/Ethnicity, Customized [Number; unit: Participants] — Ethnic population
  Participants
    Chinese | 186 | 186 | 187 | 188 | 747
    Taiwanese | 3 | 3 | 4 | 4 | 14
    Vietnamese | 10 | 10 | 9 | 10 | 39
    Indian | 35 | 37 | 35 | 37 | 144
    Filipino | 29 | 30 | 29 | 30 | 118
Pre-bronchodilator FEV1 at screening [Mean (Standard Deviation); unit: Litres] | 1.187 (0.404) | 1.192 (0.385) | 1.199 (0.415) | 1.212 (0.383) | 1.197 (0.396)
Post-bronchodilator FEV1 at screening [Mean (Standard Deviation); unit: Litres] | 1.356 (0.420) | 1.363 (0.390) | 1.366 (0.447) | 1.385 (0.408) | 1.367 (0.416)
Baseline FEV1 [Mean (Standard Deviation); unit: Litres] | 1.182 (0.415) | 1.178 (0.381) | 1.169 (0.413) | 1.184 (0.399) | 1.178 (0.402)
Smoking status [Count of Participants; unit: Participants]
  Current smoker | 84 | 85 | 86 | 85 | 340
  Former smoker | 179 | 181 | 178 | 184 | 722
Country [Count of Participants; unit: Participants]
  China | 186 | 186 | 187 | 188 | 747
  Taiwan | 3 | 3 | 4 | 4 | 14
  Vietnam | 10 | 10 | 9 | 10 | 39
  India | 35 | 37 | 35 | 37 | 144
  Philippines | 29 | 30 | 29 | 30 | 118

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in 1-hour Morning Post Forced Expiratory Volume in 1 Second (FEV1)
Description: Change from baseline in 1-hour morning post-dose FEV1 of Aclidinium bromide 400 μg/Formoterol fumarate 12 μg compared to Aclidinium bromide at Week 24.
  Baseline was defined as the average of the two FEV1 values measure prior to the administration of the first dose of the IP at randomisation visit. If one of the two values was missing, the available one was used as baseline. If both values were missing, the screening pre-bronchodilator value was used.
  Estimand is based on the while on-treatment approach, where treatment estimates are analysed while subjects are taking IP.
Time Frame: Week 24, 1-hour morning post-dose
Population: Intention-to-Treat (ITT) population: All randomised participants who took at least one dose of IP and have a baseline FEV1 measurement.
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | Placebo
Number analyzed (Participants) | 262 | 265 | 259 | 267
Litres | 0.248 (0.013) | 0.156 (0.013) | 0.138 (0.013) | -0.050 (0.013)
Statistical Analysis 1: Comparison: AB/FF 400/12 μg vs AB 400 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis — Pre-specified hierarchical sequence of testing used to adjust for multiplicity; Screening pre- and post-bronchodilator FEV1, age, baseline FEV1 as covariates; treatment, country, smoking, visit and group-by-visit as factors; Least squares mean difference = 0.092, 95% CI 2-sided [0.060 to 0.124], Standard Error of Mean 0.016

2. Primary Outcome: Change From Baseline in Morning Pre-dose (Trough) FEV1 for Aclidinium Bromide/Formoterol Fumarate
Description: Change from baseline in morning pre-dose (trough) FEV1 of Aclidinium bromide 400 μg/Formoterol fumarate 12 μg compared to Formoterol fumarate 12 μg at Week 24.
  Morning pre-dose (trough) FEV1 was defined as the average of the two FEV1 values at morning pre-dose of IP at Week 24. If one value was missing, the remaining was used as the trough value.
  Estimand is based on the while on-treatment approach, where treatment estimates are analysed while subjects are taking IP.
Time Frame: Week 24, morning pre-dose (trough)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | Placebo
Number analyzed (Participants) | 262 | 265 | 259 | 267
Litres | 0.081 (0.014) | 0.050 (0.014) | -0.004 (0.014) | -0.084 (0.014)
Statistical Analysis 1: Comparison: AB/FF 400/12 μg vs FF 12 μg; Test type: Superiority; p < 0.001, Mixed Models Analysis — Pre-specified hierarchical sequence of testing used to adjust for multiplicity; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.085, 95% CI 2-sided [0.053 to 0.117], Standard Error of Mean 0.016

3. Primary Outcome: Change From Baseline in Morning Pre-dose (Trough) FEV1 for Aclidinium Bromide
Description: Change from baseline in morning pre-dose (trough) FEV1 of Aclidinium bromide 400 μg compared to placebo at Week 24.
  Morning pre-dose (trough) FEV1 was defined as the average of the two FEV1 values at morning pre-dose of IP at Week 24. If one value was missing, the remaining was used as the trough value.
  Estimand is based on the while on-treatment approach, where treatment estimates are analysed while subjects are taking IP.
Time Frame: Week 24, morning pre-dose (trough)
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | Placebo
Number analyzed (Participants) | 262 | 265 | 259 | 267
Litres | 0.081 (0.014) | 0.050 (0.014) | -0.004 (0.014) | -0.084 (0.014)
Statistical Analysis 1: Comparison: AB 400 μg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — Pre-specified hierarchical sequence of testing used to adjust for multiplicity; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.134, 95% CI 2-sided [0.103 to 0.166], Standard Error of Mean 0.016

4. Secondary Outcome: Change From Baseline in Peak FEV1
Description: Change from baseline in peak FEV1 of Aclidinium bromide 400 μg compared to placebo at week 24.
  Peak FEV1 was the highest value recorded at Week 24 after morning IP intake.
  Estimand is based on the while on-treatment approach, where treatment estimates are analysed while subjects are taking IP.
Time Frame: Week 24, peak
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Litres
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | Placebo
Number analyzed (Participants) | 262 | 265 | 259 | 267
Litres | 0.324 (0.013) | 0.225 (0.013) | 0.191 (0.014) | 0.008 (0.014)
Statistical Analysis 1: Comparison: AB 400 μg vs Placebo; Test type: Superiority; p < 0.001, Mixed Models Analysis — Pre-specified hierarchical sequence of testing used to adjust for multiplicity; [statistical method as in outcome 1, analysis 1]; Least squares mean difference = 0.217, 95% CI 2-sided [0.184 to 0.250], Standard Error of Mean 0.017

5. Secondary Outcome: Improvements Transition Dyspnoea Index (TDI) Focal Score
Description: Improvements TDI focal score of Aclidinium bromide 400 μg/Formoterol fumarate 12 μg and Aclidinium bromide 400μg compared to placebo at week 24.
  Transition Dyspnoea Index (TDI) measures severity of breathlessness in symptomatic patients. An impairment severity score is assigned for three components: functional impairment; magnitude of task and magnitude of effort. Focal scores is derived as the sum of individual component scores. TDI focal score ranges from -9 to +9, with negative values indicating a worsening in dyspnoea, 0 showing no change from baseline and positive values associated with a post-baseline improvement.
  Estimand is based on the while on-treatment approach, where treatment estimates are analysed while subjects are taking IP.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | Placebo
Number analyzed (Participants) | 262 | 265 | 259 | 267
Units on a scale | 2.9 (0.2) | 2.6 (0.2) | 2.4 (0.2) | 2.1 (0.3)
Statistical Analysis 1: Comparison: AB/FF 400/12 μg vs Placebo; Test type: Superiority; p = 0.005, Mixed Models Analysis — Pre-specified hierarchical sequence of testing used to adjust for multiplicity; BDI, age as covariates; treatment, country, smoking, visit and group-by-visit as factors; Least squares mean difference = 0.8, 95% CI 2-sided [0.2 to 1.3], Standard Error of Mean 0.3
Statistical Analysis 2: Comparison: AB 400 μg vs Placebo; Test type: Superiority; p = 0.132, Mixed Models Analysis — Pre-specified hierarchical sequence of testing used to adjust for multiplicity; BDI, age as covariates; treatment, country, smoking, visit and group-by-visit as factors; Least squares mean difference = 0.4, 95% CI 2-sided [-0.1 to 1.0], Standard Error of Mean 0.3

6. Secondary Outcome: Change From Baseline in St Georges Respiratory Questionnaire (SGRQ) Total Score
Description: Change from baseline in SGRQ total score of Aclidinium bromide 400 μg/Formoterol fumarate 12 μg and Aclidinium bromide 400μg compared to placebo at week 24.
  St. George's Respiratory Questionnaire (SGRQ) measures the impact of COPD on overall health, daily life and perceived well-being. It is composed of 50 items split into 17 parts, from which 3 dimension scores on Symptoms, Activity and Impact are derived. A total score utilising responses to all items can also be derived to assess the overall impact of COPD on quality of life. SGRQ dimension and total scores range from 0 to 100, with higher scores indicating a worse possible health status.
  Estimand is based on the while on-treatment approach, where treatment estimates are analysed while subjects are taking IP.
Time Frame: Week 24
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: Units on a scale
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | Placebo
Number analyzed (Participants) | 262 | 265 | 259 | 267
Units on a scale | -8.7 (1.2) | -7.6 (1.2) | -7.2 (1.2) | -4.7 (1.2)
Statistical Analysis 1: Comparison: AB/FF 400/12 μg vs Placebo; Test type: Superiority; p = 0.003, Mixed Models Analysis — Pre-specified hierarchical sequence of testing used to adjust for multiplicity. P-value is nominal; Baseline SGRQ, age as covariates; treatment, country, smoking, visit and group-by-visit as factors; Least squares mean difference = -4.0, 95% CI 2-sided [-6.7 to -1.4], Standard Error of Mean 1.3
Statistical Analysis 2: Comparison: AB 400 μg vs Placebo; Test type: Superiority; p = 0.031, Mixed Models Analysis — Pre-specified hierarchical sequence of testing used to adjust for multiplicity. P-value is nominal; Baseline SGRQ, age as covariates; treatment, country, smoking, visit and group-by-visit as factors; Least squares mean difference = -2.9, 95% CI 2-sided [-5.5 to -0.3], Standard Error of Mean 1.3

ADVERSE EVENTS:
Time Frame: From time of signature of informed consent throughout the treatment period and including the follow-up period (2 weeks after last IP dose), on average 26 weeks. Only treatment-emergent AEs are reported in the tables below.
Description: An adverse event was the development of an undesirable medical condition or the deterioration of a pre-existing medical condition following or during exposure to a pharmaceutical product, whether or not considered causally related to the product. An undesirable medical condition might be symptoms, signs or the abnormal results of an investigation. The safety population was defined as all randomised patients who took at least one dose of IP.
Arm/Group | AB/FF 400/12 μg | AB 400 μg | FF 12 μg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/263 | 0/266 | 1/264 | 2/269
Serious Adverse Events (participants affected / at risk) | 19/263 | 21/266 | 26/264 | 21/269
Other Adverse Events (participants affected / at risk) | 53/263 | 44/266 | 54/264 | 55/269
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB/FF 400/12 μg (N=263) | AB 400 μg (N=266) | FF 12 μg (N=264) | Placebo (N=269)
Bronchitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cellulitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cystitis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epididymitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Gastroenteritis (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Haemorrhagic fever with renal syndrome (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Herpes zoster (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Infective exacerbation of chronic obstructive airways disease (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Keratitis viral (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Laryngopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Lower respiratory tract infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 2 (2) | 3 (3) | 5 (5) | 4 (4)
Postoperative wound infection (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Sepsis (Infections and infestations) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Benign neoplasm of adrenal gland (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Benign neoplasm of skin (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Bladder papilloma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Rectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Lymphadenitis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Thrombocytosis (Blood and lymphatic system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Basal ganglia haemorrhage (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cerebral arteriosclerosis (Nervous system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Cerebral haemorrhage (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Cluster headache (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Spondylitic myelopathy (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Transient ischaemic attack (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cataract (Eye disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Iridocyclitis (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vertigo (Ear and labyrinth disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Acute coronary syndrome (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Acute myocardial infarction (Cardiac disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Angina unstable (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Cardiac failure congestive (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Myocardial infarction (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Myocardial ischaemia (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 9 (10) | 6 (6) | 10 (10) | 7 (7)
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pulmonary mass (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Gastric polyps (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gastritis erosive (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Inguinal hernia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Large intestine polyp (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hepatic function abnormal (Hepatobiliary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Intervertebral disc protrusion (Musculoskeletal and connective tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Acute kidney injury (Renal and urinary disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Chronic kidney disease (Renal and urinary disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Death (General disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Foot fracture (Injury, poisoning and procedural complications) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tendon rupture (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | AB/FF 400/12 μg (N=263) | AB 400 μg (N=266) | FF 12 μg (N=264) | Placebo (N=269)
Upper respiratory tract infection (Infections and infestations) | 31 (32) | 25 (28) | 24 (27) | 24 (28)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 25 (33) | 21 (28) | 33 (44) | 35 (43)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2021-07-08): https://cdn.clinicaltrials.gov/large-docs/97/NCT03022097/Prot_000.pdf
  • Statistical Analysis Plan (2022-05-06): https://cdn.clinicaltrials.gov/large-docs/97/NCT03022097/SAP_001.pdf